CLINICAL TRIAL: NCT00025532
Title: A Pre-Phase I Biodistribution Study Of hCC^CH2 Labeled With 131 Iodine In Patients With Gastrointestinal Adenocarcinomas
Brief Title: Radiolabeled Monoclonal Antibody Therapy in Treating Patients With Gastrointestinal Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068971; UCSF-H11156-18101-02; UCSF-00455; NCI-T97-0054
Record Dates: First submitted 2001-10-11; First posted 2003-11-21 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer; Esophageal Cancer; Gastric Cancer; Pancreatic Cancer
Keywords: stage III colon cancer; stage IV colon cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage III pancreatic cancer; recurrent pancreatic cancer; stage III rectal cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus; adenocarcinoma of the colon; adenocarcinoma of the rectum; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Colorectal Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Colonic Neoplasms; Rectal Neoplasms; Adenocarcinoma Of Esophagus

INTERVENTIONS:
Other: iodine I 131 monoclonal antibody CC49-deltaCH2

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and deliver tumor-killing substances to them without harming normal cells. This may be an effective treatment for gastrointestinal cancer.

PURPOSE: Phase I trial to study the effectiveness of radiolabeled monoclonal antibody therapy in treating patients who have gastrointestinal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the biodistribution and biokinetics of iodine I 131-labeled monoclonal antibody CC49-delta CH2 in patients with gastrointestinal adenocarcinoma. II. Determine the human anti-human monoclonal antibody response in patients treated with this drug.

OUTLINE: Patients receive iodine I 131-labeled monoclonal antibody CC49-delta CH2 (131I MOAB CC49-delta CH2) IV over 5-10 minutes on day 0. Patients also receive unlabeled monoclonal antibody CC49-delta CH2 IV over 5 minutes followed by 131I MOAB CC49-delta CH2 IV over 5-10 minutes on day 28. Patients are followed weekly for 4 months and then every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the esophagus, stomach, pancreas, colon, or rectum More than 30% positively immunoreactive to monoclonal antibody CC49 in the metastatic or primary lesion OR TAG-72 antigen serum level greater than 15 Measurable or evaluable unresectable or metastatic disease by CT scan

PATIENT CHARACTERISTICS: Age: 19 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC greater than 3,500/mm3 Platelet count greater than 150,000/mm3 Hemoglobin greater than 10 g/dL Hepatic: Bilirubin less than 2.0 mg/dL ALT and AST less than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present) PTT less than 37.0 seconds INR less than 2.0 Renal: Creatinine less than 2.0 mg/dL Other: No known allergy to murine immunoglobulin No iodine allergy No concurrent illness that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Must be ambulatory and able to comply with study schedule

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior murine immunoglobulin Chemotherapy: Prior or concurrent chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy allowed Surgery: See Disease Characteristics

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2001-04

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A. Tempero, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Cancer Center and Cancer Research Institute, San Francisco, California, United States